CLINICAL TRIAL: NCT03484377
Title: Measuring Cortical Dynamics of Inhibitory Control Before, During and After Transcranial Direct Current Stimulation (tDCS)
Brief Title: Cortical Dynamics of Inhibitory Control: A Concurrent tDCS-MEG Study
Acronym: CDIC-tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Najat Khalifa (Other Government)
Collaborators: Medical Research Council (Other Government); University of Nottingham (Other)
Responsible Party: Sponsor-Investigator, Najat Khalifa, Associate Professor, Nottinghamshire Healthcare NHS Trust
Organization: Nottinghamshire Healthcare NHS Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CiC2017051; 199-1801 (Other: Research Ethics - University of Nottingham)
Record Dates: First submitted 2018-03-14; First posted 2018-03-30 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Impulsive Behavior
MeSH Terms: conditions — Impulsive Behavior | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Concurrent tDCS-MEG parallel arms single-blinded experimental design (right anodal v sham tDCS).
Who Masked: Participant
Masking Description: Participants will be randomly allocated, using a computer generated code, to receive either anodal tDCS or sham. For sham stimulation, the current will be delivered only in the first 10 seconds, after which the stimulation will cease but with the electrodes still in place throughout the session
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anodal tDCS (Experimental): The anodal tDCS electrode will be placed over the area corresponding to the right DLPFC (F4 of the EEG10-20 international system). The anodal tDCS condition will use a constant current of 2mA, delivered via gradual increase and decrease over 10 seconds at the onset and offset of stimulation (current ramps), respectively.
  Interventions: Device: Anodal tDCS
- Sham tDCS (Sham Comparator): The sham (cathodal) electrode will be placed over the left supraorbital ridge. The current will be delivered only in the first 10 seconds, after which the stimulation will cease but with the electrodes still in place throughout the session.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS — The experimental condition will use a constant current of 2mA for 20 minutes, delivered via gradual increase and decrease over 10 seconds at the onset and offset of stimulation (current ramps), respectively.
  Arms: Anodal tDCS
Device: Sham tDCS — The anodal electrode will be placed over the supreorbital ridge. The current will be delivered only in the first 10 seconds, after which the stimulation will cease but with the electrodes still in place throughout the session. The session will last for 20 minutes.
  Arms: Sham tDCS

SUMMARY:
This study aims to use concurrent Transcranial Direct Current Stimulation (tDCS) and Magnetoencephalography (MEG) with measures of impulsivity to examine the neurobiological underpinnings of rapid response impulsivity (RRI) and how these can be modified using tDCS in healthy subjects.

DETAILED DESCRIPTION:
Concurrent tDCS-MEG parallel arms single-blinded experimental design (right anodal v sham tDCS) will be employed in this study. The study will be conducted at the University of Nottingham, using a sample of student volunteers. This study aims to examine the influence of anodal tDCS on beta-band and alpha-band oscillatory activities, using an anti-saccade task administered before, during and after tDCS stimulation. It can potentially help understand the neurobiological mechanisms underpinning rapid response impulsivity and how these can be influenced by tDCS.

The research hypotheses are that (i) a generalised mechanism for top-down inhibitory control will play a vital role, whereby prefrontal beta-band activity initiates alpha-band activity for functional inhibition over the frontal eye fields and other areas in the neurocircuitry involved in RRI; (ii) anodal tDCS (as opposed to sham) delivered over the right DLPFC will enhance this mechanism; and (iii) there will be no significant correlations between measures of self-report impulsivity and performance on the anti-saccade task and measures of oscillatory activity.

ELIGIBILITY:
Inclusion Criteria:

* University students and staff
* Aged 18-40

Exclusion Criteria:

* Individuals with epilepsy and other neurological conditions, history of significant head injury, substance misuse, major mental disorder and those receiving psychotropic medication.
* Contraindications to use of Magnetic Resonance (pacemakers, metal implants, aneurysm clips)
* Pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Total number of correct anti-saccade (AS) trials | Change from baseline after 20 minutes of tDCS
  A measure of rapid response impulsivity (inhibitory control)

SECONDARY OUTCOMES:
Total number of correct pro-saccade (PS) trials | Change from baseline after 20 minutes of tDCS
  A behavioral measure of rapid response impulsivity (inhibitory control)
Saccade latency for anti-saccade (AS) trials | Change from baseline after 20 minutes of tDCS
  A behavioral measure of rapid response impulsivity (inhibitory control)
Saccade latency for pro-saccade (PS) trials | Change from baseline after 20 minutes of tDCS
  A behavioral measure of rapid response impulsivity (inhibitory control)
Total Scores on the UPPS+P Impulsive Behaviour Scale | Baseline
  A self-report measure of impulsivity
Alpha and Beta band activity | Change from baseline after 20 minutes of tDCS
  A Cortical measure of inhibitory control recorded using Magnetoencephalography (MEG). MEG is a brain imaging technique.

OTHER OUTCOMES:
Alpha and Beta band activity | During 20 minutes of tDCS stimulation
  Evaluation of mechanism of action of tDCS using MEG data

CONTACTS AND LOCATIONS:
Overall Officials: Najat Khalifa, DM, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03484377/Prot_000.pdf